CLINICAL TRIAL: NCT06066762
Title: Monitoring of Argatroban Anticoagulant Therapy in Patients With Acute Suspected Heparin-induced Thrombocytopenia: French Multicenter Study
Brief Title: Argatroban Monitoring in Acute Suspected Heparin-induced Thrombocytopenia.
Acronym: TIH-FM
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231085
Record Dates: First submitted 2023-09-28; First posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Heparin-induced Thrombocytopenia
Keywords: thrombocytopenia; argatroban; fibrin monomers
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Nature of samples: plasma from a tube of citrated blood
  * Quantity/volume of samples taken: between 3 and 5 ml per collection time and according to the practice of the participating centres
  * Quantity/volume of samples kept for research purposes: between 2 to 3 plasma aliquots of 400 μl / patient corresponding to the samples taken as part of the care and during the follow-up of the participant - Storage conditions: - 80°C
  * Identification of aliquots: registration of the unique and project-specific identification number + Acronym of the project
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Heparin-induced thrombocytopenia (HIT) is a rare but potentially serious complication of heparin therapy. , argatroban is the alternative anticoagulant of choice in patients with suspected HIT and renal impairment, high bleeding risk or risk of invasive surgery/gesture. Despite its increasing use in these fragile patients, methods for biological monitoring of argatroban's anticoagulant activity are heterogeneous, and neither the therapeutic zone nor the modalities for argatroban dosage adjustment are clearly defined, particularly in patients in the acute phase of thrombosis.

Soluble fibrin monomers (FM) indirectly reflect thrombin generation in vivo. This marker could thus represent a new strategy for monitoring the anticoagulant activity of argatroban. However, the effect of argatroban anticoagulation on FM levels remains unknown.

In a preliminary retrospective study carried out at Bichat hospital, we showed that FM levels could therefore be an early marker of the efficacy of argatroban treatment in patients with suspected HIT.In order to confirm these results, we will include patients with clinico-biological suspicion of HIT and receiving argatroban treatment.

Ten French laboratories will participate in this study. All plasmas collected will be from samples taken only in the context of care.

This prospective study will determine whether the daily monitoring of FM is beneficial for the management of patients treated with argatroban.

DETAILED DESCRIPTION:
The study plan to set up a multicenter biobank of plasmas from patients treated with argatroban for suspected HIT in 10 French hematology laboratories (Dijon, Nantes, Tours, Lille, Bordeaux, Nancy, St Etienne, Lariboisière, Rennes, Bichat) that have agreed to participate in this study and have expertise in the management of these patients. All centers adapted the dose of argatroban to its activity, using a test to measure its concentration (TTd or ECT). Some centers adapt the argatroban dose in addition to the anti-IIa activity on FMs, while others do not.

Patient recruitment :

Patients will be recruited over a 1-year period starting in end of 2023. All patients with suspected HIT for whom argatroban therapy is initiated will be included, including patients on ECMO. Plasma from tube ends will be frozen (minimum 2 aliquots of 400 µL) in each center. FMs will be measured daily in centers adapting argatroban dosage to FMs. In other centers, FMs will be measured either daily on fresh plasma or a posteriori on frozen plasmas.

Sampling procedure :

All samples are taken as part of the treatment. No additional tubes will be taken specifically for research purposes.

* D0: A sample will be taken just before starting argatroban, until D-2 before starting argatroban treatment.
* D1: A sample will be taken at least 4 hours after the start of treatment
* D2 to D8: A sample will be taken daily at least 4 hours after any dose change (if applicable)
* D10 and D14: A sample will be taken at least 4 hours after any dose change (if applicable).

In each center: daily plasma storage (2x400 µl minimum) at -80°C.

Analyses performed :

* on fresh whole blood/plasma: blood cell count, aPTT, fibrinogen, anti-IIa activity, D-dimer for all centers. FM for centers1 2 3 (n=50 patients)
* on fresh or frozen plasma: FM for centers 4 5 6 7 8 9 10 (n=50 patients)

ELIGIBILITY:
Inclusion Criteria:

* patients suspected of having HIT in any department, including ECMO in the 10 centers
* patient starting a treatment with argatroban.
* major patients

Exclusion Criteria:

* Minor patients
* Patient under legal protection (guardianship or curatorship)
* Patient objecting to re-use of data and samples

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient with suspected heparin-induced thrombocytopenia and for whom Argatroban is prescribed as part of the treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Adaptation of the argatroban dose on FM (fibrin monomers) to allow better dose adjustment of Argatroban in patients with suspected HIT | 12 days
  The study will help determine whether this dose adjustment of Argatroban on FM allows an earlier rise of platelets as well as a decrease in thrombotic and/or hemorrhagic events compared to centers that do not use FM.

SECONDARY OUTCOMES:
Determine the therapeutic zone for argatroban, which is not clearly defined to date, based on the following main criteria: FM negativation, correction of thrombocytopenia, absence of thrombotic and hemorrhagic events. | 12 days

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Ajzenberg, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Bichat-Claude Bernard, Paris, France